CLINICAL TRIAL: NCT03062449
Title: A Phase IIa Proof of Concept, Randomized, Double-blind, Placebo-controlled Study of the Effects of L-serine on Early Stage Alzheimer's Disease Patients
Brief Title: Phase IIa L-serine Trial for eAD
Acronym: LSPI-2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stability of investigational product could not be established.
Sponsor: Aleksandra Stark (Other)
Collaborators: Brain Chemistry Labs (Other)
Responsible Party: Sponsor-Investigator, Aleksandra Stark, MD, Assistant Professor of Neurology, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D16180
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Alzheimer Disease
Keywords: L-Serine, Alzheimer's Disease, AD, Memory,
MeSH Terms: conditions — Alzheimer Disease | interventions — Serine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- L-Serine Gummy Arm (Active Comparator): L-serine will be presented in gummies containing 1g serine each. Subjects randomized into the L-serine arm will take 15 grams of L-Serine (15 gummies containing 1g of L-serine) orally twice daily for 246 days after the initial ascending dose period to confirm tolerability of the dose.
  Interventions: Drug: L-Serine
- Placebo Gummy Arm (Placebo Comparator): Placebo gummies containing no L-serine will be packaged in the same manner as that of the L-Serine gummy arm and be given to patients to take two times a day.
  Interventions: Other: Placebo Gummy

INTERVENTIONS:
Drug: L-Serine — Gummy containing L serine dose
  Arms: L-Serine Gummy Arm
Other: Placebo Gummy — Gummy with no dosing of L Serine
  Arms: Placebo Gummy Arm

SUMMARY:
This is a Phase IIa, randomized, double-blind, placebo controlled trial. Subjects for participation in this study will be identified by the Investigator based on their Clinical Dementia Rating score which will be completed as part of standard practice. Patients meeting the criteria for early Alzheimer's disease will be considered for study participation, with the Investigator taking the additional inclusion/exclusion criteria into consideration. Up to 40 subjects will be enrolled. Subjects participating in the study will be randomized to receive either gummies containing L-Serine or placebo gummies, with the Investigator and study staff blinded to the group assignments.

DETAILED DESCRIPTION:
L-serine (C3H7NO3; 105.09 g/mol; synonym (S)-2-amino-3-hydroxypropanoic acid) is a naturally-occurring dietary amino acid. It is abundant in soy products, some edible seaweeds, sweet potatoes, eggs, and meat. Since some L-serine is produced by astrocytes in the brain, it is considered a non-essential amino acid. L-serine is directly involved in the biosynthesis of purines, pyrimidines, and other amino acids. Serine residues are found in most proteins and within proteins function as a site for phosphorylation.

L-serine is considered as GRAS (generally recognized as safe) by the FDA and has been approved as a normal food additive under CFR172.320. It is widely sold as a dietary supplement. A pilot study of L-serine supplementation of 14 patients with hereditary sensory neuropathy has been published, and subsequent trial is on-going (ClinicalTrials.gov identifier NCT01733407). The authors did not report adverse effects at doses of 400mg/kg/day, which for an average American of 75.5kg is about 30 grams, the dose which we propose to use in this study.

L-serine will be administered orally through gummies. Each gummy contains 1 g L-serine (treatment) and will be packaged in a foil packet containing 15 pieces to be taken both morning and evening for nine months. The placebo will be a gummy containing no L-serine, packaged and taken in the same manner. In order to assess tolerability in patients, we have designed a 4 week dose ramp-up. We will monitor side-effects and amino acid balances in blood samples in the early Alzheimer's Disease patients during a dose ramp-up period. If a patient cannot tolerate the full dose of gummies, they will remain in the study taking a total of 1 package of gummies split into two time periods within the day. The same ramp-up schedule and procedures will be observed for both placebo and L-serine patients. Patients will be assessed at baseline, 3 months, 6 months, and 9 months.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of early stage Alzheimer's disease as scored by the ClinicalDementia Rating Scale score of 0.5 -1.0 within the 6 months prior to study enrollment.
2. Participants able to provide informed consent.
3. Participants taking NMDA receptor antagonist medications or acetylcholinesterase inhibitor medications must be on a stable dose of these medications for at least 30 days prior to enrolling in this clinical trial.
4. Participants able to consume study gummy chews throughout the course of the clinical trial.

Exclusion Criteria:

1. Diagnosis or previous history of ischemic stroke, astrocytoma, meningioma or oligodendroma.
2. Diagnosis or previous history of any other comorbid diagnosis of neurodegenerative disease including amyotrophic lateral sclerosis, Parkinson's disease, Lewy Body Disease, Pick's Disease, Huntington's Disease, or Progressive Supra Nuclear Palsy.
3. Undergoing any chemotherapy or radiation therapy for any tumor or carcinoma.
4. Diagnosis or previous history of type I or type II diabetes. Potential subjects with no history of diabetes will be referred to their PCP for a hemoglobin A1C test if they have not had one in the year prior to enrollment.
5. Diagnosis or previous history of psychiatric illness that in the investigator's opinion would affect the subject's ability to successfully participate in the study.
6. In the Investigator's opinion, subject would be unable to successfully participate in the study for any reason.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra C Stark, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was placed on voluntary hold by the institution prior to study completion. Upon review of the stability data of the investigational agent provided by the product's manufacturer, the FDA IND Sponsor-Investigator (PI) and institutional officials determined that the available information was unsatisfactory. No reportable study outcome data are available as determined by the institution and Sponsor-Investigator (PI) because the stability of the investigational product cannot be verified.
Pre-assignment Details: Study participants are grouped for the participant flow. The study was closed by the Sponsor-Investigator and institution prior to study completion because the stability of the investigational product could not be verified.
Period: Overall Study
Arm/Group | L-Serine Gummy Arm | Placebo Gummy Arm
Started | 16 | 13
Completed Treatment | 10 | 12
Completed (Completed all follow-up) | 9 | 12
Not Completed | 7 | 1
Not completed — Withdrawal by Subject | 7 | 1

BASELINE CHARACTERISTICS:
Population: All study participants are grouped for the baseline measure and reported for all participants collectively. The study was closed by the PI and institution prior to study completion because the stability of the investigational product could not be verified.
Groups:
- Total: Total of all reporting groups
Arm/Group | L-serine Gummy Arm | Placebo Gummy Arm | Total
Number analyzed (Participants) | 16 | 13 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 7
  >=65 years | 11 | 11 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 13 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 13 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in Score on the Montreal Cognitive Assessment Assessment Evaluation
Description: Cognitive Assessment will be performed and score obtained at clinical trial visits. The Montreal Cognitive Assessment or The MoCA Test is a highly sensitive tool for early detection of mild cognitive impairment. The assessment evaluates eight domains of cognitive functions, including visuospatial and executive function, naming, memory, attention, language, abstraction, and orientation. Scores on the MoCA range from 0 to 30. A score less than 26 is considered as mild cognitive impairment. Higher values represent a better outcome.
Time Frame: Baseline, 6 Months, 9 Months
Population: Investigational agent stability data provided by product's manufacturer was determined to be unsatisfactory by the Sponsor-Investigator (PI) and institutional officials. The study was closed by the PI and institution prior to study completion. Data are potentially invalid due to the inadequate stability testing performed by the manufacturer, as the sponsor-investigator is unable to confirm that the investigational product remained stable over time. No reportable study outcome data are available.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | L-Serine Gummy Arm | Placebo Gummy Arm
Number analyzed (Participants) | 16 | 13
score on a scale
  Baseline | 20.625 [16 to 25] | 22.923 [14 to 30]
  6 Months: number analyzed (Participants) | 13 | 11
  6 Months | 19.846 [12 to 24] | 21.909 [15 to 28]
  9 Months: number analyzed (Participants) | 10 | 10
  9 Months | 20.3 [14 to 27] | 21.5 [13 to 29]

2. Secondary Outcome: Change in Plasma Biomarker Levels.
Description: Levels of biomarkers related to cognitive status will be assessed in plasma that was collected at clinical trial visits.
Time Frame: Baseline, 6 Months, 9 months
Population: Investigational agent stability data provided by product's manufacturer was determined to be unsatisfactory by the Sponsor-Investigator (PI) and institutional officials. The study was closed by the PI and institution prior to study completion. Data are potentially invalid due to the inadequate stability testing performed by the manufacturer, as the sponsor-investigator is unable to confirm that the investigational product remained stable over time. The biomarker data does not exist.
Arm/Group | L-Serine Gummy Arm | Placebo Gummy Arm
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Relationship Between Montreal Cognitive Assessment Score and Plasma Biomarker Levels
Description: Disease status biomarker levels will be assessed in plasma at trial visits. Montreal Cognitive Assessment testing will be performed and scored at each visit.
Time Frame: Baseline, 6 Months, 9 months
Population: as for outcome 2
Arm/Group | L-Serine Gummy Arm | Placebo Gummy Arm
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Self-reported L-serine Tolerability
Description: Each participant will report tolerability on a scale of 1 to 10 (1 = poor and 10 = excellent). This assessment was completed at the end of participation via a phone calls 4 weeks after visit 4.
Time Frame: 4 weeks (+/- 2 weeks) after visit 4 (week 36 +/- 2 weeks)
Population: Investigational agent stability data provided by product's manufacturer was determined to be unsatisfactory by Sponsor-Investigator (PI) and institutional officials. The study was closed by PI and institution prior to study completion. Data are potentially invalid due to inadequate stability testing performed by the manufacturer, as PI is unable to confirm that investigational product remained stable over time. Only 10 participants from L-serine and 7 from placebo group completed the assessment.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | L-Serine Gummy Arm | Placebo Gummy Arm
Number analyzed (Participants) | 10 | 7
units on a scale | 8 [1 to 10] | 8 [1 to 10]

5. Other Pre Specified Outcome: Number of Clinically Significant Lab Values for Complete Blood Count, Liver Function Test, Basic Metabolic Panel Measures.
Description: Health check labs will be collected from every participant at each clinical trial visit. clinically significant lab values will be identified for complete blood count, liver function test, and basic metabolic panel measures.
Time Frame: Baseline, 3 Months, 6 Months, 9 months
Population: Investigational agent stability data provided by product's manufacturer was determined to be unsatisfactory by the Sponsor-Investigator (PI) and institutional officials. Data are potentially invalid due to the inadequate stability testing performed by the manufacturer, as the sponsor-investigator is unable to confirm that the investigational product remained stable over time. The number of participants analyzed decreased over time due to participants withdrawing or being withdrawn by the PI.
Measure: Number; unit: # of clinically significant lab values
Arm/Group | L-Serine Gummy Arm | Placebo Gummy Arm
Number analyzed (Participants) | 16 | 13
# of clinically significant lab values
  Baseline | 0 | 0
  3 Months: number analyzed (Participants) | 14 | 12
  3 Months | 0 | 0
  6 Months: number analyzed (Participants) | 13 | 10
  6 Months | 0 | 0
  9 Months: number analyzed (Participants) | 10 | 10
  9 Months | 0 | 0

ADVERSE EVENTS:
Time Frame: Investigational agent stability data provided by product's manufacturer was determined to be unsatisfactory by the Sponsor-Investigator (PI) and institutional officials. Study was closed by the PI and institution prior to study completion. Data are potentially invalid due to inadequate stability testing performed by the manufacturer; the sponsor-investigator is unable to confirm that investigational product remained stable overtime. Adverse event data were collected over approximately 4 months.
Description: Due to the inability to confirm adherence with the study treatment (Gummy Bears) by the subjects enrolled in the study, the attribution of any adverse events (including serious events) to study treatment is not possible. Thus, adverse events are being reported in aggregate.
Groups:
- L-Serine: Gummy Arm: L-serine will be presented in gummies containing 1g serine each. Subjects randomized into the L-serine arm will take 15 grams of L-Serine (15 gummies containing 1g of L-serine) orally twice daily for 246 days after the initial ascending dose period to confirm tolerability of the dose.
  L-Serine: Gummy containing L serine dose
Arm/Group | L-Serine: Gummy Arm | Placebo Gummy Arm
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/16 | 2/13
Other Adverse Events (participants affected / at risk) | 16/16 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-Serine: Gummy Arm (N=16) | Placebo Gummy Arm (N=13)
chest pain (General disorders) | 1 (1) | 0 (0) — chest pain
gastroenteritis (Gastrointestinal disorders) | 0 (0) | 2 (3) — gastroenteritis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-Serine: Gummy Arm (N=16) | Placebo Gummy Arm (N=13)
movement disorder (Nervous system disorders) | 1 (2) | 1 (1) — abnormal movement
skin lesion or rash (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) — injury
sleep disturbance (Psychiatric disorders) | 3 (5) | 0 (0) — sleep disruption
weight gain (Investigations) | 3 (4) | 3 (3) — weight gain
cataract extraction (Eye disorders) | 2 (2) | 1 (1) — surgery
syncope (Nervous system disorders) | 1 (1) | 0 (0) — syncope
bradycardia (Cardiac disorders) | 1 (1) | 0 (0) — bradycardia
diarrhea (Gastrointestinal disorders) | 5 (6) | 2 (2) — diarrhea
cognitive decline (Nervous system disorders) | 3 (3) | 7 (8) — cognitive decline
weight loss (Investigations) | 2 (2) | 2 (2) — weight loss
anxiety (Psychiatric disorders) | 1 (1) | 1 (1) — anxiety
dog bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — injury
tic bite (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) — injury
potential overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — over dose
atrophy of hands (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — atrophy
pneumonia (Infections and infestations) | 0 (0) | 1 (1) — pneumonia
leg edema (Vascular disorders) | 1 (1) | 1 (1) — edema
pulmonary vascular congestion (Vascular disorders) | 0 (0) | 1 — vascular congestion
cellulitis (Infections and infestations) | 0 (0) | 2 (2) — cellulitis
recurrent major depressive disorder (Psychiatric disorders) | 0 (0) | 1 (1) — depression
taste change (Nervous system disorders) | 1 (1) | 0 (0) — taste change
reduced appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) — reduced appetite
nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) — nausea
gas (Gastrointestinal disorders) | 1 (2) | 2 (2) — gas
reduced platelets (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — reduced platelets
change in bowel habits (Gastrointestinal disorders) | 1 (1) | 0 (0) — change in bowel habits
hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — hiccups
headache (Nervous system disorders) | 1 (1) | 1 (1) — headache
upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) — URI
fatigue (General disorders) | 0 (0) | 1 (1) — fatigue
peripheral neuropathy (Nervous system disorders) | 0 (0) | 1 (1) — neuropathy
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — abdominal pain
worsening vision secondary to left cataract (Eye disorders) | 1 (1) | 0 (0) — visual decline
dental procedure (Surgical and medical procedures) | 1 (1) | 0 (0) — procedure
blood pressure elevation (Vascular disorders) | 0 (0) | 1 (1) — hypertension
focal pain above left breast (Reproductive system and breast disorders) | 0 (0) | 1 (1) — pain
right hearing impairment (Ear and labyrinth disorders) | 0 (0) | 1 (1) — hearing loss
hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) — hypothyroidism
hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — hyperlipidemia
cold (General disorders) | 1 (1) | 1 (1) — cold
puncture wound left foot (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — injury
irritability (Psychiatric disorders) | 2 (2) | 2 (2) — agitation
lightheadedness (Nervous system disorders) | 1 (1) | 0 (0) — lightheadedness
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — nasal congestion
flashing lights at night (Eye disorders) | 1 (1) | 0 (0) — flashing lights
feeling sped up (Psychiatric disorders) | 1 (1) | 0 (0) — anxiety
right ear infection (Infections and infestations) | 1 (1) | 0 (0) — infection
gout (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) — gout
lack of motivation (Psychiatric disorders) | 0 (0) | 1 (1) — lack of motivation
soft tissue injury due to fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) — injury
arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — arthritis
increased restlessness (Psychiatric disorders) | 0 (0) | 1 (1) — agitation
hot flashes (Vascular disorders) | 0 (0) | 1 (1) — hot flashes
falls, no injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — falls

LIMITATIONS AND CAVEATS:
The Sponsor-Investigator (PI) and institutional officials determined that the available investigational agent stability data of provided by the product's manufacturer was unsatisfactory. The study was closed by the PI and institution prior to study completion. Data are potentially invalid due to the inadequate stability testing performed by the manufacturer, as the sponsor-investigator is unable to confirm that the investigational product remained stable over time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT03062449/Prot_SAP_000.pdf